CLINICAL TRIAL: NCT02023671
Title: IMMUNOPHENOTYPE ROLE IN THE EVALUATION OF CLINICAL RESPONSE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Benedetto Bruno, MD, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: MM-EMD-2013
Record Dates: First submitted 2013-12-24; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Myeloma; Post Allografting
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study proposed by SSCVD Allogeneic Stem Cells of this Hospital provides for the collection of a series composed of patients with multiple myeloma undergoing allogeneic stem cell transplants at our center in the period 2000-2011.

This collection is carried out with retrospective investigation , through the review of paper and electronic records and data cards already collected as part of clinical trials conducted by our own Division and approved by the Ethics Committee of Management.

The purpose of data collection is particularly retrospective analysis of the incidence of extramedullary relapse , the response in flow cytometry immunophenotypic and clinical response of the disease , will also be taken into consideration for overall survival ( OS) , event-free survival (EFS) , the cumulative incidence of treatment-related mortality and graft- versus-host disease ( GVHD ), acute and chronic.

The data were processed in a completely anonymous and as provided by law. The results of the study will not result in any diagnostic or therapeutic intervention on patients still alive.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with multiple myeloma undergoing allogeneic stem cell transplantation in the period 2000-2011 at the University Transplant Center of the Division of Hematology.

Were taken into account both donor transplants voluntary blood relative.

Exclusion Criteria:

Patients who died early after allogeneic transplantation (<3 months) in which has not been evaluated disease status.

In the evaluation of the response of immunophenotypic disease were excluded from the analysis of bone marrow aspirate samples with low cellularity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
Event free survival | 5 years